CLINICAL TRIAL: NCT04462224
Title: Creation of Home-based Asthma Real-World Measures With Mobile Health (CHARM) Study
Brief Title: Creation of Home-based Asthma Real-World Measures With Mobile Health Study
Acronym: CHARM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Jewish Health (Other)
Responsible Party: Sponsor
Other Study IDs: HS-3476
Record Dates: First submitted 2020-05-14; First posted 2020-07-08 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Asthma
Keywords: Asthma; Asthma control; Biologics; Biologic therapy; Quality of life; Biologic therapies; Mobile health; Moderate-to-Severe; Asthma exacerbation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Four novel biologic therapies (benralizumab, dupilumab, mepolizumab, reslizumab) have been recently approved for moderate-to-severe, eosinophilic or oral steroid-dependent asthma. The efficacy and safety of these therapies have been determined primarily by randomized clinical trials that compared annualized rates of significant asthma exacerbations (SAEs), lung function changes, and standardized symptom survey score changes in therapy-treated subjects in comparison to placebo matched controls. Yet, there is increasing interest to assess the efficacy, health benefits, and safety in medical therapies using real-world evidence (RWE). Further, home monitoring of asthma using mobile health (mHealth) technology may help scientists develop new and more sensitive indicators of asthma control that could improve clinical care. The hypothesis is that real world evidence, collected at home using several mobile health technologies, will help determine the efficacy, health benefits, and side effects of these therapies.

Objectives

1. Assess real-world evidence (RWE) indicators of worsening and improving asthma. Scientists will measure steps per day, duration and vigor of exercise per day, sleep quality, and the number of awakenings per night using Fitbit activity trackers. Scientists will measure symptoms using once-monthly custom survey delivered to participant smartphones via Twilio. Rescue medication use and adherence to maintenance medications may be measured using digital inhaler devices. Adherence to biologic use using HealthBeacon smart sharps containers may be measured. Measures collected will be correlated to patient-reported significant asthma exacerbations (SAEs), lung function (FEV1), and the asthma control test (ACT) collected in clinic every 3 months.
2. Use RWE to determine responses to biologic therapies. Scientists will combine at-home and clinic data to determine responses to biologics.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of uncontrolled or difficult-to-treat asthma, defined as 1 course of systemic corticosteroids (e.g. oral prednisone) in the last 12 months
* OR -
* An asthma control test (ACT) score less than or equal to 19 despite regular use of inhaled corticosteroids (ICS) therapy (at least 176 mcg of fluticasone/day or the equivalent)
* Participants will need access to a smartphone (As of January 2018, ~ 80% of U.S. adults owned a smartphone (Mobile Fact Sheet, 2018))

Exclusion Criteria:

* Active smoking
* Any significant comorbid conditions that could inadvertently interfere with study results (i.e. any terminal illness, cancer, HIV, end-stage renal disease, congestive heart failure, severe autoimmune disease or inflammatory bowel disease)
* Conditions that require bursts of oral corticosteroids
* Other significant lung diseases (cystic fibrosis, pulmonary hypertension, interstitial lung disease, pulmonary fibrosis among others) to be determined by the investigators.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with uncontrolled, moderate-to-severe asthma.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Asthma Control Test | Baseline to 24 or 52 weeks
  Standardized asthma symptom survey

SECONDARY OUTCOMES:
Change From Baseline in Significant asthma exacerbations | Baseline and Week 24 (Phase 1) or Week 52 (Phase 2)
  A protocol-defined asthma exacerbation was defined as worsening of asthma symptoms requiring treatment with systemic corticosteroids for 3 or more days; for patients receiving long-term oral corticosteroids, an exacerbation was a 20 mg or more increase in average daily dose of oral prednisone (or a similar dose of another systemic corticosteroid). The rate of protocol-defined asthma exacerbations, normalized by subject-time at risk and computed over the 24 observation or 52-week treatment period in each treatment group.
Change From Baseline in Lung Function | Baseline and Week 24 (Phase 1) or Week 52 (Phase 2)
  FEV1 % predicted pre- and post-bronchodilator FEV1 absolute (L) pre- and post-bronchodilator FVC % predicted pre- and post-bronchodilator FVC absolute (L) pre- and post-bronchodilator Bronchodilator response: % change in FEV1 after bronchodilator FEV1/FVC ratio: absolute and % predicted. Aggregated measure: significant vs non significant bronchodilator reversibility. Significant reversibility defined as greater than or equal to 12% and 200mL increase in FEV1 or FVC
Change From Baseline in Number of Puffs per Day of Beta Agonist Rescue Medication | Baseline and Week 24 (Phase 1) or Week 52 (Phase 2)
  Number of inhalations per day averaged out over the study's duration Number of inhalations per night per month averaged out over the study's duration
Change From Baseline in Adherence of Inhaled Corticosteroids | Baseline and Week 24 (Phase 1) or Week 52 (Phase 2)
  Doses taken/doses prescribed average out over the study's duration
Change From Baseline in Adherence of Biologics | Baseline and Week 24 (Phase 1) or Week 52 (Phase 2)
  Doses taken/doses prescribed average out over the study's duration
Change From Baseline in Steps Per Day | Baseline and Week 24 (Phase 1) or Week 52 (Phase 2)
  Steps per day average out over study's duration
Change From Baseline in Duration and Intensity of Exercise Per Day | Baseline and Week 24 (Phase 1) or Week 52 (Phase 2)
  Minutes exercise per day average out over study's duration Minutes exercise/day x average heart rate during the exercise
Change From Baseline in Duration of Interrupted Sleep per Night | Baseline and Week 24 (Phase 1) or Week 52 (Phase 2)
  Hours of uninterrupted sleep as recorded by Fitbit device
Change From Baseline in Number of Awakenings per Night | Baseline and Week 24 (Phase 1) or Week 52 (Phase 2)
  Number of awakenings per night and/or early morning awakenings as a composite score, as recorded by Fitbit
Change From Baseline in the Monthly Symptom Questionnaire Scores | Baseline and Week 24 (Phase 1) or Week 52 (Phase 2)
  Each answer will be scored 1-10 points, depending on the answer, and added to create a survey score. Higher scores indicate poorer asthma control.

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States